CLINICAL TRIAL: NCT06503536
Title: REAL-world Patient characterISTICs, Treatment Pattern, Clinical Outcomes, and Healthcare Resource Utilization in Chinese Patients Receiving Upadacitinib for Atopic Dermatitis: A Retrospective Chart Review Study
Brief Title: A Study to Assess Treatment Patterns, Clinical Outcomes, and Healthcare Resource Utilization in Chinese Participants Receiving Upadacitinib for Atopic Dermatitis (AD) Through Chart Review
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: H24-962
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic Dermatitis (AD); Upadacitinib
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants with Atopic Dermatitis (AD) undergo chart review up to180 days after initiating upadacitinib.

SUMMARY:
Atopic Dermatitis (AD) is a common, chronic, and flaring systemic inflammatory skin disorder characterized by intensely pruritic and distressing skin eruptions. This study will assess treatment patterns, treatment outcomes, healthcare resource utilization in Chinese participants receiving Upadacitinib for Atopic Dermatitis (AD) undergoing chart review.

ELIGIBILITY:
Inclusion Criteria:

* Participants with at least one primary diagnosis of atopic dermatitis with ICD-10 code of L20.900 [atopic dermatitis, unspecified] or physician-confirmed atopic dermatitis documentation within the study period
* Participants with at least one documented health record of upadacitinib prescription that has a primary diagnosis of atopic dermatitis within the study period
* Participants with at least one atopic dermatitis severity measures (i.e., EASI) in the follow-up period including up to 6 months after the index date

Exclusion Criteria:

• Participants who did not fulfill the inclusion criteria will be excluded

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Atopic Dermatitis (AD) receiving Upadacitinib undergoing chart review in China
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who achieve a composite endpoint post-index score of Eczema Area and Severity Index (EASI) < =7 | Up to 3 months
  Eczema Area and Severity Index (EASI): Clear=0, Almost clear=0.1-1.0, Mild=1.1-7.0, Moderate=7.1-21.0, Severe=21.1-50.0, Very severe=50.1-72.0
Number of participants who achieve a composite endpoint post-index score of Investigator's Global Assessment (IGA) × Body Surface Area (BSA) < = 30 | Up to 3 months
  Investigator's Global Assessment (IGA) × Body Surface Area (BSA): Mild=0-30, Moderate=30.1-130, Severe=130.1-400

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Huashan Hospital affiliated to Fudan University /ID# 268259, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=H24-962